CLINICAL TRIAL: NCT01956396
Title: Phase I of Study of Safety and Efficacy of the PrePex Device for MC Programs in Zimbabwe
Brief Title: Evaluation of Safety and Efficacy of the PrePexTM Device for Rapid Scale up of Adult MC Programs in Zimbabwe
Acronym: ZW-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ministry of Health and Child Welfare, Zimbabwe (Other)
Responsible Party: Principal Investigator, Prof. Mufuta Tshimanga, Public Health Physician, Department of Community Medicine, University of Zimbabwe, Ministry of Health and Child Welfare, Zimbabwe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MRCZ/A/1628 Safety Study
Record Dates: First submitted 2012-09-19; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Circumcision Adult; HIV CDC Category B2; HIV Infections
Keywords: male circumcision; HIV; Zimbabwe
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: PrePex™ device (Experimental): Adult male circumcision by the PrePex™ device
  Interventions: Device: PrePex™ device

INTERVENTIONS:
Device: PrePex™ device — PrePex™ device for adult male circumcision. The non-surgical PrePex™ device with No Injected Anesthesia

SUMMARY:
The protocol, approved by the Medical Research Council, was issued to assess the safety and efficacy of the non-surgical device for applying it to the national scale up of adult male circumcision in Zimbabwe

DETAILED DESCRIPTION:
Models show that to have the highest impact on the HIV epidemic, circumcision of up to 80% of men in high prevalence countries, where MC rates are low, needs to be achieved (UNAIDS 2009; Manicaland HIV/STD Prevention Project, 2008; Bollinger, et al, 2009). Hallett and colleagues in 2008 showed that for Zimbabwe specifically, HIV incidence could be reduced between 25% to 35% if about 50% of men are circumcised. All modelings conducted show that MC programs must be part of a comprehensive HIV prevention package as MC alone will not tip the HIV epidemic into a terminal decline.

The PrePex Device offers hope for rapid scale up of adult male circumcision in resource limited settings.

Once the safety and efficacy have been established, it is important to conduct operations research to determine how best to implement both device and surgical circumcisions in the national program. Thus, the Zimbabwe MOHCW is planning a three phase trial in order to determine the safety of the PrePexTM device, its performance and the ease of use in an implementation roll out.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 30 years
* Uncircumcised
* Wants to be circumcised
* Agrees to be circumcised by any of the study methods,PrePex or Surgical as appropriate
* HIV sero-negative
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse and to keep caution not to directly rub the cut area if masturbating, for 8 weeks post removal (9 weeks total)
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 8 weeks post removal (9 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits
* Agrees to stay overnight at the Hospital in order to follow pain measurements in the first 16 hours

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* HIV sero-positive
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality
* Uncontrolled diabetes
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits
* Refusal to take HIV test.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The Safety and Efficacy of the PrePex Device for adult male circumcision in Zimbabwe | 8 week post-procedure follow up appointment and examination
  Outcome measures include:
  Clinical adverse events and device-related incidents

SECONDARY OUTCOMES:
Evaluating the procedure duration | 8 week post-procedure follow up appointment and examination
  The total procedure and preparation time of the PrePex™ device circumcision procedure
Evaluating the pain at key time points | 8 week post-procedure follow up appointment and examination
  Pain assessment at key time points using Visual Analog Scale (VAS)
Evaluating the discomfort during daily activities | 8 week post-procedure follow up appointment and examination
  using questionnaires
Evaluating the compliance during use (with follow-up) | 8 week post-procedure follow up appointment and examination
  compliance during use (with follow-up)using questionnaires
Evaluating the procedure acceptability by Doctors | 8 week post-procedure follow up appointment and examination
  procedure acceptability by Doctors using questionnaires
Glans fully exposed | 8 week post-procedure follow up appointment and examination
Evaluating time to complete healing | 8 week post-procedure follow up appointment and examination
  time to complete healing using wound assessment
Evaluating the cosmetic results | 8 week post-procedure follow up appointment and examination
Procedure acceptability by Nurses | 8 week post-procedure follow up appointment and examination
  Procedure acceptability by Nurses using questionnaires
Satisfaction by subjects | 8 week post-procedure follow up appointment and examination
  Satisfaction by subjects
Satisfaction by providers | 8 week post-procedure follow up appointment and examination
  using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gwinji, MBChB, MPH, Principal Investigator — PS- MoHCW
Locations (1):
- Znfpc Spilhaus Center, Harare, Zimbabwe

REFERENCES:
- See also: MRCZ — http://www.mrcz.org.zw/